CLINICAL TRIAL: NCT02710097
Title: Ethanol and Cannabinoid Effects on Simulated Driving and Related Cognition: Sub-Study II
Acronym: THC-ETOH-II
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1501015208.B
Record Dates: First submitted 2016-03-10; First posted 2016-03-16 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cannabis; Alcohol Effect; Driving Under the Influence of Alcohol and Other Drugs
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active THC and Placebo Ethanol (Experimental)
  Interventions: Drug: Active inhaled cannabis; Drug: Placebo
- Active THC and Active Ethanol (Experimental)
  Interventions: Drug: Active inhaled cannabis; Drug: Active Oral Ethanol
- Placebo THC and Active Ethanol (Experimental)
  Interventions: Drug: Active Oral Ethanol; Drug: Placebo
- Placebo THC and Placebo Ethanol (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active inhaled cannabis — ~450 mg of active cannabis, which is roughly equivalent to smoking 1/4 of a marijuana cigarette, or "joint". Administered over 20 minutes via a vaporizer.
  Arms: Active THC and Active Ethanol; Active THC and Placebo Ethanol
Drug: Placebo — Approximately 4 drinks of orange juice or ginger ale covered with a trace amount of ethanol on the surface, each administered over approximately 10 minutes.
  Arms: Active THC and Placebo Ethanol; Placebo THC and Placebo Ethanol
Drug: Active Oral Ethanol — 0.4 g/kg ethanol in orange juice or ginger ale to reach a target BrAC of approximately 0.04%. This dose is equivalent to approximately 2 standard drinks over 1 hour. Approximately 4 drinks, each administered over approximately 10 minutes.
  Arms: Active THC and Active Ethanol; Placebo THC and Active Ethanol
Drug: Placebo — No active cannabinoids. Administered over 20 minutes via a vaporizer.
  Arms: Placebo THC and Active Ethanol; Placebo THC and Placebo Ethanol

SUMMARY:
The overarching goal of this study is to characterize the effects of ethanol and cannabinoids on simulated driving and related cognition.

DETAILED DESCRIPTION:
To study the effects of oral ethanol (target BAC of ~0.04g/dl; equivalent to consuming approximately 2 drinks over 1 hour) and vaporized cannabis (~450 mg cannabis plant material at a THC concentration of ~1.7%; roughly equivalent to smoking approximately 1/4 of a marijuana cigarette, or "joint") on driving.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 21 to 55 years of age (extremes included).
* Occasional current cannabis users.
* Experience with drinking 2 or more standard drinks of alcohol at least once in lifetime.
* Able to provide informed consent.

Exclusion Criteria:

* Cannabis naïve.
* Alcohol naïve.
* Positive pregnancy screen
* Hearing deficits.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Road Tracking Error | baseline, +20, +50, +120, +180 mins after start of alcohol administration

SECONDARY OUTCOMES:
Biphasic Alcohol Effects Scale (BAES) | baseline, +20, +50, +120, +180, +240 mins after start of alcohol administration
  A scale designed to assess the stimulant and sedative effects associated with alcohol intoxication
Visual Analog Scale (VAS) | baseline, +20, +50, +120, +180, +240 mins after start of alcohol administration
  Feeling states associated with alcohol and cannabis intoxication will be measured using this self-report scale of feeling states.
Cognitive Test Battery | +40 mins after start of alcohol administration
  Several computer tasks will be administered to assess alcohol and THC effects on driving related cognition, including:
  visual vigilance, visual motor function, attention and working memory, and processing speed.
Willingness to Drive Scale | baseline, +20, +50, +120, +180, +240 mins after start of alcohol administration
  Subjects will be asked to rate their willingness to drive at their current state in the context of various scenarios including willingness to drive from testing facility to a number of destinations that are different driving distances.
Number of Joints Scale | baseline, +20, +50, +120, +180, +240 mins after start of alcohol administration
  Subjects will be asked to rate the number of standard joints that they believe they have been administered.
Number of Drinks Scale | baseline, +20, +50, +120, +180, +240 mins after start of alcohol administration
  Subjects will be asked to rate the number of standard drinks that they believe they have been administered.

CONTACTS AND LOCATIONS:
Locations (1):
- Biological Studies Unit, VA Connecticut Healthcare System, West Haven, Connecticut, United States